CLINICAL TRIAL: NCT04466371
Title: Perceptions of Undergraduate Students and Teaching Staff on Online Teaching and Learning in the Wake of COVID-19 Pandemic in an Egyptian Private University: A Cross-Sectional Study
Brief Title: Perceptions of Undergraduate Students and Teaching Staff on Online Teaching
Status: Suspended | Type: Observational
Why Stopped: Administrative problems
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Other Study IDs: PUB 1114005
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-01

CONDITIONS: Covid19
Keywords: Online learning; Teaching methods; COVID-19 knowledge and perceptions
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MIU students and staff members: All students and staff members in MIU
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — A questionnaire to assess satisfaction with online learning and knowledge about COVID-19

SUMMARY:
Spread of COVID-19 in the world has led to a shift in teaching and learning techniques to online methods in order to prevent transmission of the disease. Misr International University (MIU) has an established online learning system that has been used together with face-to-face classes. The aim of this study is to assess and compare the satisfaction and perceptions of full-time teaching staff and undergraduate students regarding online learning during COVID-19 crisis.

DETAILED DESCRIPTION:
Statement of the problem: Spread of COVID-19 in the world has led to a shift in teaching and learning techniques to online methods in order to prevent transmission of the disease. Misr International University (MIU) has an established online learning system that has been used together with face-to-face classes. However, shifting all courses in all the faculties to the online mode is a new experience that needs to be assessed to allow for future improvement plans.

Aim: To assess and compare the satisfaction and perceptions of full-time teaching staff and undergraduate students regarding online learning during COVID-19 crisis.

Method: An online anonymous questionnaire will be distributed to all Misr International University (MIU) students and staff members. The total number of students is 8679 and the total number of staff members regardless of their academic title is 530. The questionnaire will be validated by three experts and piloting will be performed on a sample of participants. The questionnaire consists of five sections: Demographics, satisfaction with online teaching and learning methods, knowledge, and perception of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* All MIU undergraduate students and full-time staff members

Exclusion Criteria:

* Students or full-time staff members who will not respond to the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All undergraduate MIU students and staff members who respond to the questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 9209 (Estimated)
Dates: Start 2027-07-15 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with online learning | 1 month
  Assess level of satisfaction with online learning using a questionnaire

SECONDARY OUTCOMES:
Knowledge about COVID-19 crisis | 1 month
  Assess level of knowledge about COVID-19 using a questionnaire
Perception of COVID-19 crisis | 1 month
  Assess level of perception of COVID-19 crisis using a questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral & Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Questionnaire and results can be shared

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Bryan, A. & Volchenkova, Kseniya.. Blended Learning: Definition, Models, Implications for Higher Education. 2016;8: 24-30. doi:10.14529/ped160204.
- [Background] Pei L, Wu H. Does online learning work better than offline learning in undergraduate medical education? A systematic review and meta-analysis. Med Educ Online. 2019 Dec;24(1):1666538. doi: 10.1080/10872981.2019.1666538. PMID 31526248
- [Background] Mohammadi, Neda & Ghorbani, Vahid & Hamidi, Farideh.. Effects of e-learning on Language Learning. Procedia CS. 2011;3: 464-468. doi:10.1016/j.procs.2010.12.078.
- [Background] ABC of Content Validation and Content Validity Index Calculation.
- See also: Middle East Respiratory Syndrome (MERS) Global Summary and Assessment of Risk (2019). World Health Organization (WHO). — http://www.who.int/emergencies/mers-cov/en/
- See also: WHO announces COVID-19 Outbreak a Pandemic. World Health Organization Regional Office for Europe (2020). — https://www.euro.who.int/en/health-topics/health-emergencies/coronavirus-covid-19/news/news/2020/3/who-announces-covid-19-outbreak-a-pandemic
- See also: ESTELAMI, H. (2013). Frontiers of distance learning in business education — http://site.ebrary.com/id/10928490
- See also: International Association of Universities Global Survey Report on The Impact of COVID-19 on Higher Education Around the World (2020) — https://www.iau-aiu.net/IMG/pdf/iau_covid19_and_he_survey_report_final_may_2020.pdf